CLINICAL TRIAL: NCT04124679
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Sleep After Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAES and sleep
Record Dates: First submitted 2019-10-08; First posted 2019-10-11 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Transcutaneous Electrical Acupoint Stimulation; Thoracoscopic Surgery; Postoperative Sleep Quality

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAES group (Experimental): In TEAS group, an experienced acupuncturist performed 30 minutes of TEAS treatment at the HT7 (Shenmen) and Neiguan (PC6) acupoints on bilateral side, which were identiﬁed in accordance with the TCM anatomic localizations on the first night before surgery by a stimulator (Hwato Electronic Acupuncture Treatment Instrument, model no.: SDZ-II; Suzhou Medical Appliances Co. Ltd, Suzhou, China). And after surgery, ST36 (Zusanli) and LI4 (Hegu) acupoints were added for the effect of relieving postoperative complications. 30 minutes of TEAS treatment was also performed on bilateral side by an experienced acupuncturist at the Neiguan (PC6), HT7 (Shenmen), ST36 (Zusanli) and LI4 (Hegu) acupoints on the first three nights after surgery
  Interventions: Other: Transcutaneous Electrical Acupoint Stimulation
- Control group (No Intervention): Patients in the control group were attached the gel electrodes at the sham acupoints

INTERVENTIONS:
Other: Transcutaneous Electrical Acupoint Stimulation — patients received Transcutaneous Electrical Acupoint Stimulation for 30 mins on the acupoints
  Arms: TAES group

SUMMARY:
General anesthesia is a medically induced state of low reactivity consciousness which is similar to natural sleep.Some studies found that general anesthesia as an independent risk factor could result in a desynchronization of the circadian time structure and cause postoperative sleep disorders characterized by reduced rapid eye movement (REM) and slow wave sleep (SWS),which have signiﬁcant deleterious impacts on postoperative outcomes, such as postoperative fatigue, severe anxiety and depression, emotional detachment and delirium, and even pain sensitivity or postoperative pain of patients.Acupuncture can regulate plant nerve activity by increasing slow-wave sleep time to improve sleep quality.The results of polysomnography monitoring showed that the sleep latency, total sleep time, awakening index and sleep quality were all significant improved after acupuncture treatment.And transcutaneous electrical acupoint stimulation（TAES） works by stimulating Shu yu acupoints, which is more convenient than the normal electric acupuncture. The purpose of this paper is to study the effect of TAES on sleep after thoracoscopic surgery

DETAILED DESCRIPTION:
In TEAS group, an experienced acupuncturist performed 30 minutes of TEAS treatment at the HT7 (Shenmen) and Neiguan (PC6) acupoints on bilateral side, which were identiﬁed in accordance with the TCM anatomic localizations on the first night before surgery by a stimulator (Hwato Electronic Acupuncture Treatment Instrument, model no.: SDZ-II; Suzhou Medical Appliances Co. Ltd, Suzhou, China). And after surgery, ST36 (Zusanli) and LI4 (Hegu) acupoints were added for the effect of relieving postoperative complications. 30 minutes of TEAS treatment was also performed on bilateral side by an experienced acupuncturist at the Neiguan (PC6), HT7 (Shenmen), ST36 (Zusanli) and LI4 (Hegu) acupoints on the first three nights after surgery. The TEAS was standardized before each treatment and was set at 2/10 HZ, which has been documented as the most effective frequency. The optimal intensity is from 6 to 15mA, which was adjusted according to individual maximum tolerance to maintain a slight twitching of the regional muscles. Patients in the control group were attached the gel electrodes at the sham acupoints. The acupuncture points were to be stimulated by microcurrents generated by a special electrical device, which the patients may only experience a mild electric current sensation or nothing at all.

ELIGIBILITY:
Inclusion Criteria:

* ASA ( American Society of Anesthesiologists):I-II
* age for 18-75 years

Exclusion Criteria:

* History of central nervous system and mental illness
* use of sedatives or antidepressants
* infection or wound at the percutaneous acupuncture point
* unwilling to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
sleep quality tested by sleep monitor of the second night before the operation | second night before the surgery
  using sleep monitor to test the sleep quality on second night before the operation, analyze sleep quality according to each percentage of sleep stage.
sleep quality tested by sleep monitor of the first night before the operation | the first night before surgery
  using sleep monitor to test the sleep quality on first night before the operation, analyze sleep quality according to each percentage of sleep stage..
sleep quality tested by sleep monitor of the first night after the operation | the first night after the operation
  using sleep monitor to test the sleep quality on the first night after the operation,analyze sleep quality according to each percentage of sleep stage.
sleep quality of the tested by sleep monitor on the third night after the operation | the third night after the operation
  using sleep monitor to test the sleep quality on the third night after the operation,analyze sleep quality according to each percentage of sleep stage.

SECONDARY OUTCOMES:
subjective sleep quality: Athens Insomnia Scale | one night before the operation and the first and third night after the operation
  using the Athens Insomnia Scale to test the subjective sleep quality of patients. The range were from 0-3. Total score < 4 means sleep well; total score =6 means suspicious of insomnia; total score > 6 means insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Junchao h Zhu, Study Director — Shengjing Hospital
Locations (1):
- Shengjing hospital of China Medical university, Shenyang, Liaoning, China